CLINICAL TRIAL: NCT01093443
Title: Administration of a GnRH Antagonist During 3 Days at Initiation of the Cycle: Impact on the Stimulation in IVF/ICSI
Brief Title: Gonadotropin-releasing Hormone (GnRH) Antagonist During 3 Days
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Paul Devroey, Universitair Ziekenhuis Brussel
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009/196
Record Dates: First submitted 2010-03-24; First posted 2010-03-25 (Estimated); Last update posted 2010-10-11 (Estimated); Status verified 2009-11

CONDITIONS: Infertility
Keywords: IVF; ICSI; GnRH antagonist; pretreatment
MeSH Terms: conditions — Infertility | interventions — Ovulation Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Placebo Comparator): Patients undergo a standard treatment with a classical GnRH antagonist protocol.
  Interventions: Drug: ovarian stimulation
- B (Active Comparator): Before undergoing a standard protocol for ovarian stimulation, patients in this group receive a pretreatment with GnRH antagonists during 3 consecutive days
  Interventions: Drug: ovarian stimulation

INTERVENTIONS:
Drug: ovarian stimulation — rFSH with GnRH antagonists
  Arms: A
Drug: ovarian stimulation — GnRH antagonist, rFSH, GnRH antagonist
  Arms: B

SUMMARY:
In this prospective study, the investigators would like to show whether ovarian stimulation with pretreatment of a GnRH antagonist during 3 consecutive days at initiation of the cycle, is possible.

DETAILED DESCRIPTION:
A recently accepted study demonstrated that raised progesterone levels can be normalized through administration of a GnRH antagonist during three subsequent days prior to the start of gonadotropin stimulation in a GnRH antagonist protocol. This regimen, after normalisation of the progesterone value, allows controlled ovarian hyperstimulation (COH). Since this regimen is valid in case of elevated progesterone, GnRH antagonists pretreatment may prove to be a valid tool for scheduling IVF treatment in patients with normal progesterone values on day 2 of the cycle. In this prospective randomised trial, the investigators study the impact of administration of a GnRH antagonist during 3 consecutive days at initiation of the cycle.

ELIGIBILITY:
Inclusion Criteria:

* < 39 years old on day of randomisation
* FSH < 12 (in the early follicular phase)
* Normal ultrasound scan, i.e. presence of both ovaries, without evidence of abnormality within 6 months prior to randomisation.
* Regular menstrual cycles of 21-35 days, presumed to be ovulatory.
* BMI between 18 and 29 (both inclusive)
* 1st or 2nd trial
* IVF or ICSI
* Randomisation at out-patient clinic

Exclusion Criteria:

* ≥ 39 years old on day of randomisation
* Endometriosis ≥ grade 3
* PCOS

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Endocrine profile | up to 9 months
  The purpose is to assess the endocrine profile in each treatment group

SECONDARY OUTCOMES:
Pregnancy rate | up to 9 months
  The purpose is to study the pregnancy rate in each treatment group

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Brussel, Jette, Brussels Capital, Belgium